CLINICAL TRIAL: NCT06352151
Title: Comparison of the Effects of Orofacial Therapy and Therapeutic Yoga on Swallowing, Sleeping Habits and Quality of Life in Children With Down Syndrome
Brief Title: Effects of Orofacial Therapy and Therapeutic Yoga in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, YASEMİN KOTEVOĞLU, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-041
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-08

CONDITIONS: Down Syndrome
Keywords: Myofunctional Therapy; Yoga; Down Syndrome; Quality of Life; Swallowing; Sleep Habits
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Grup: Routine Physiotherapy Group (Experimental): Children with Down Syndrome receive routine physiotherapy treatment in special education centers.
  Interventions: Other: Routine Physiotherapy Group
- 2.Group: Orofacial Treatment Group (Experimental): The orofacial treatment group receives therapeutic orofacial treatment in addition to routine physiotherapy treatment. For orofacial therapy, sessions will be conducted twice a week for eight weeks, lasting 30-45 minutes, totaling 16 sessions.
  Interventions: Other: Orofacial Treatment Group
- 3.Group: Therapeutic Yoga Group (Experimental): The therapeutic yoga group receives therapeutic yoga treatment and routine physiotherapy treatment. Sixteen sessions were planned twice a week for eight weeks, each 30-45 minutes.
  Interventions: Other: Therapeutic Yoga Group

INTERVENTIONS:
Other: Routine Physiotherapy Group — Children with Down syndrome who receive routine physical therapy treatment in special education centers will undergo evaluation after eight weeks of treatment, followed by a control evaluation after 12 weeks.
  Arms: 1. Grup: Routine Physiotherapy Group
Other: Orofacial Treatment Group — The orofacial treatment group receives therapeutic orofacial treatment in addition to routine physiotherapy treatment. Each week, one or two target exercises will be taught to the child with Down syndrome, and the exercises will gradually increase throughout the process. Parental involvement will be encouraged during the treatment to ensure active participation in therapy.
  The goals of the therapy are as follows:
  First Goal: Nasal hygiene and Sleep hygiene education
  Second Goal: Nasal Breathing Exercise Training
  Third Goal: Creating Awareness of Tongue Resting Position
  Fourth Goal: Creating Lip Position Awareness - Lip Exercises
  Goal Five: Chewing Muscle Exercises
  Sixth Goal: Strengthening the Soft Palate
  Seventh Goal: Reshaping Correct Swallowing
  Arms: 2.Group: Orofacial Treatment Group
Other: Therapeutic Yoga Group — The therapeutic yoga group receives therapeutic yoga treatment and routine physiotherapy treatment. Children with Down syndrome will be given yoga exercises suitable for their age.
  Arms: 3.Group: Therapeutic Yoga Group

SUMMARY:
The study aims to compare the effects of orofacial therapy and therapeutic yoga on swallowing, sleep habits, and quality of life in children with Down syndrome.

DETAILED DESCRIPTION:
At special education and rehabilitation centers, children diagnosed with Down syndrome will undergo initial assessment, and those meeting the inclusion criteria will be included in the study following parental voluntary consent.

Measurement assessments will be conducted three times: before therapy, after therapy (at week 8), and at a follow-up at week 12. To ensure a fair and unbiased distribution, children participating in the study will be randomly assigned to their respective groups using a sealed envelope method, a widely accepted and transparent randomization technique.

1. Grup: Routine Physiotherapy (PT) Group - Receiving routine physiotherapy treatment.

   Children who receive routine physiotherapy treatment in special education centers will be evaluated at the end of the 8th session following the treatment. After 12 weeks, the control will be in the form of an evaluation.
2. Grup: Orofacial Therapy + Routine PT Group - Receiving orofacial therapy and routine physiotherapy treatment.

   For the orofacial therapy, sessions will be held twice a week for eight weeks, with each session lasting 30-45 minutes, totaling 16 sessions. This structured and intensive therapy schedule is designed to provide a comprehensive evaluation of the therapy's effectiveness. Secondary evaluations will be conducted following the 8th treatment session, and a follow-up evaluation will be performed after 12 weeks.
3. Grup: Therapeutic Yoga Group + Routine PT Group - Receiving therapeutic yoga and routine physiotherapy treatments.

The therapeutic yoga group at special education centers will also meet twice weekly for eight weeks, each lasting 30-45 minutes, for 16 sessions. Secondary evaluations will be conducted following the 8th treatment session, and a follow-up evaluation will be performed after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Age between 5 and 12 years old
* Scoring 4 or higher on the pEAT-10 questionnaire
* Obtained parental consent form
* Ability of the child to cooperate

Exclusion Criteria:

* Conditions that would impede assessment or communication (such as cognitive problems, psychiatric issues, etc.).
* Children who have undergone any surgery related to orofacial structures and/or received orthodontic treatment.
* Those with a history of trauma (whiplash injury, condylar trauma, fractures).
* Children who have received orofacial-related physical therapy treatment within less than 6 months.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
The Pediatric Functional Independence Measure | Baseline, 8 weeks,12 weeks
  The Pediatric Functional Independence Measure (WeeFIM): The WeeFIM consists of 18 items across 6 separate domains. These domains include self-care, sphincter control, transfers, mobility, communication, and social-cognitive evaluations. When answering the items in the WeeFIM sections, scoring is based on whether assistance is needed during the activity, and whether any assistive devices are required. The WeeFIM scale yields scores ranging from a minimum of 18 to a maximum of 126 points.
Pediatric Eating Assessment Tool-10 | Baseline, 8 weeks, 12 weeks
  The Pediatric Eating Assessment Tool-10 (p-EAT-10) is a scale consisting of 10 items used to screen the severity of dysphagia symptoms. Each item is scored from 0 to 4 (0=No problem and 4=Severe Problem). Normative data indicate that a p-EAT-10 score of 4 or higher indicates a risk of swallowing disorder, with higher scores indicating more severe dysphagia symptoms.
Children's Sleep Habits Questionnaire | Baseline, 8 weeks,12 weeks
  The Children's Sleep Habits Questionnaire (CSHQ) form contains 33 items, including 8 subscales. The CSHQ assesses the following subscales: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night waking, parasomnias, sleep-disordered breathing, and daytime sleepiness. The scale is filled out retrospectively by parents. A total score of 41 points is considered the cutoff point for the CSHQ, and scores above this threshold indicate that children are experiencing clinically significant sleep problems.
The Health-Related Quality of Life Scale-KIDSCREEN-27 | Baseline, 8 weeks,12 weeks
  The Health-Related Quality of Life Scale-KIDSCREEN-27 form is drawn from the KIDSCREEN-52 and consists of 27 questions and 5 dimensions. The dimensions of KIDSCREEN-27 include physical well-being (5 items), psychological well-being (7 items), autonomy and relationships with parents (7 items), social support and peers (4 items), and school environment (4 items). In all KIDSCREEN questionnaires, items have a 5-point Likert-type response scale (never, seldom, sometimes, often, always). An increase in score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)